CLINICAL TRIAL: NCT05945524
Title: Analysis of the Resistance and Sensitivity Mechanisms to Teclistamab by Focusing on Single Immune Cell Examination
Acronym: ResisTec
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: RC31/23/0278
Record Dates: First submitted 2023-05-16; First posted 2023-07-14 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Multiple Myeloma
Keywords: Teclistamab; Resistance; Immune Cell
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Analysis of bone marrow (Experimental): Analysis of bone marrow in patients initiated treatment by Teclistamab for 18 cycles
  Interventions: Other: Bone marrow sampling

INTERVENTIONS:
Other: Bone marrow sampling — Bone marrow sampling collected at 12 weeks after initiation treatment (day 1 cycle 4)

SUMMARY:
The aim of this study is to discover the immune and oncogenomic features that distinguish patients who respond to teclistamab from patients who are primarily resistant. Moreover, phenotypic and genotypic characteristics that occur with secondary resistance to teclistamab will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* With multiple myeloma
* Who receive Teclistamab
* Consent form signed

Exclusion Criteria:

* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-09-28 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Response to teclistamab at 12 weeks | at day 1 Cycle 4 (each cycle is 28 days)
  response according to International Myeloma Working Group criteria

CONTACTS AND LOCATIONS:
Overall Officials: Hervé AVET LOISEAU, MD, PhD, Principal Investigator — University Hospital, Toulouse
Locations (18):
- France (18):
  - CHU d'Amiens, Amiens, France
  - CHU de Caen, Caen, France
  - Polyclinique du Parc Drevon, Dijon, France
  - CH Annecy Genevois, Epagny Metz- Tessy, France
  - CHU de Lille, Lille, France
  - Centre Léon Bérard, Lyon, France
  - CHU de Montpellier, Montpellier, France
  - Hôpital Saint-Louis, Paris, France
  - Hôpital Saint-Antoine, Paris, France
  - Hôpital Necker, Paris, France
  - CHU de Bordeaux, Pessac, France
  - CHU de Lyon, Pierre-Bénite, France
  - CHU de Poitiers, Poitiers, France
  - CHU de Rennes, Rennes, France
  - CH Saint-Etienne, Saint-Priest-en-Jarez, France
  - CHU de Toulouse, Toulouse, France
  - CHU de Tours, Tours, France
  - CHRU Nancy, Vandœuvre-lès-Nancy, France

IPD SHARING:
Plan to Share IPD: No